CLINICAL TRIAL: NCT02407158
Title: A Pilot Study to Explore Alternative Methods for Verifying Endotracheal Tube Repositioning in the Surgical Intensive Care Unit
Brief Title: Pilot Study for Verifying Endotracheal Tube Repositioning Using Ultrasound
Status: Terminated | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1502015336
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Endotracheal Tube Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SonarMed Airwave Device — Measure the concordance of chest x-ray and the Airwave device for measuring the change of position of an endotracheal tube.

SUMMARY:
The investigators will compare the response to oral endotracheal tube repositioning as measured by chest x-ray and measured by the air-wave device.

DETAILED DESCRIPTION:
Patients This prospective, non-randomized observational study will be conducted in the Surgical Intensive Care Unit (SICU) at Yale-New Haven Hospital. As this is a pilot study to determine the accuracy and precision of the SonarMed® AirWave™ monitor, the investigators have based our projected enrollment population to complete the study within one year. Intubated patients in the SICU requiring ETT repositioning will be identified by SICU clinicians (attending physicians, residents, respiratory therapists, and registered nurses). Based on manufacturer restrictions, patients with ETTs smaller than 6.5mm and larger than 9mm, double lumen ETTs, and those patients receiving Heliox therapy will be excluded from this study.

Study Procedures Once the patient is identified by a member of the clinical care team, this will be communicated to the research team.

A member of the research team will verify eligibility for the study, and then place the sensor and monitoring device into the airway circuit. The monitor is placed at the end of the endotracheal tube, in-line with the ventilator circuit.

Once the required distance for ETT repositioning is prescribed, the respiratory therapist will move the ETT based on the positioning at the incisors. This is standard practice. The device readings will be recorded pre- and post-repositioning. The therapist will be blinded to the device readings. The readings taken from the AirWave monitor are for research purposes only, and will not be considered when making clinical care decisions. Following repositioning, it is standard practice to obtain a follow up chest X-ray for confirmation of tube position within a two hour window. The same head positioning, noted on the original X-ray, will be maintained for the follow up X-ray. Device readings will also be taken at the time of the follow up X-ray. If the tube is to be further repositioned based on the decisions of the SICU team the device will be left in place until such time as the tube position has been fully optimized by the SICU team.

The ETT movement recorded by the AirWave™ monitoring device will be compared with the position change indicated on the chest X-ray. Once this has been completed, the monitor will be discontinued and removed.

For this study, additional data will be recorded: name, hospital record number, age, height, weight, gender, race, prior medical history, reason for SICU admission, reason for intubation, complications due to mechanical ventilation, days on mechanical ventilation (number of days prior to repositioning procedure and total number of days), length of stay, vital signs pre- and post-repositioning, including oxygen saturation, FiO2, and any peri-procedural vital sign abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Intubated patients in the SICU requiring ETT repositioning will be identified by SICU clinicians.

Exclusion Criteria:

* Based on manufacturer restrictions, patients with ETTs smaller than 6.5mm and larger than 9mm, double lumen ETTs, and those patients receiving Heliox therapy will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated patients in the SICU requiring ETT repositioning will be identified by SICU clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Correlation between tube position measured by chest x-ray and the Air-Wave Device | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Davis, MD, MBA, Study Chair — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States